CLINICAL TRIAL: NCT05798104
Title: Improving Patient Knowledge and Confidence in Specialty Biologic Self-administration Through Collaborative Nurse-pharmacist Counseling
Brief Title: Collaborative Nurse-pharmacist Counseling for Self-administered Biologics
Acronym: COLLAB
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: research is not clinically appropriate at this time due to competing demands and patient care
Sponsor: Tonia Carr (Other)
Responsible Party: Sponsor-Investigator, Tonia Carr, Nurse Manager, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 80874
Record Dates: First submitted 2023-03-17; First posted 2023-04-04 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Medication Adherence; Medication Nonadherence; Adverse Drug Event
MeSH Terms: conditions — Medication Adherence; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Collaborative nurse-pharmacist counseling (Experimental): Collaborative nurse-pharmacist counseling - At the interventional appointment, study participants will first complete a modified Okere-Reiner pre-survey assessing patient perceptions of confidence and knowledge in their biologic therapy. Subsequently, a pharmacist will perform a refresher medication counseling, detailing indication, dosing, storage, and side effects. Upon completion of this counseling, an infusion nurse will then provide education demonstrating proper self-administration to the patient. The patient will then self-administer the medication with coaching and direct observation from the nurse. Afterwards, the patient will complete the Okere-Reiner post-survey to determine the effectiveness of the counseling session at improving perceived confidence and knowledge. Patients will complete both the pre-and post-surveys with direct entry to REDCap on an institution iPad during the study intervention visit.
  Interventions: Behavioral: Collaborative nurse-pharmacist counseling

INTERVENTIONS:
Behavioral: Collaborative nurse-pharmacist counseling — At the interventional appointment, study participants will first complete a modified Okere-Reiner pre-survey assessing patient perceptions of confidence and knowledge in their biologic therapy. Subsequently, a pharmacist will perform a refresher medication counseling, detailing indication, dosing, storage, and side effects. Upon completion of this counseling, an infusion nurse will then provide education demonstrating proper self-administration to the patient. The patient will then self-administer the medication with coaching and direct observation from the nurse. Afterwards, the patient will complete the Okere-Reiner post-survey to determine the effectiveness of the counseling session at improving perceived confidence and knowledge. Patients will complete both the pre-and post-surveys with direct entry to REDCap on an institution iPad during the study intervention visit.

SUMMARY:
The goal of this clinical trial is to learn if nurse-pharmacist counseling can improve patient knowledge and confidence and prevent side effects in patients who start a biologic medication in-office and later continue the medication at home. The main question it aims to answer are:

• Does nurse-pharmacist counseling improve patient-reported knowledge and confidence in biologic self-treatment when moving from in-office to at-home administration?

Participants will attend a brief counseling session in office and respond to a pre-counseling and post-counseling survey to look at medication knowledge and confidence. Participants will be contacted at three months after the survey to ask if they had any side effects related to their biologic medicine. Data will be collected from the participant's medical record at the study institution for up to six months after the study counseling session.

ELIGIBILITY:
Inclusion Criteria:

* Referred to University of Kentucky Specialty and Infusion Services for clinic-administration of a biologic medication
* Biologic medication is omalizumab, risankizumab-rzaa or ustekinumab
* Medication administration will be transitioned to self-administration

Exclusion Criteria:

* Less than 18 years of age
* have previously received the qualifying biologic at another institution
* non-English speaking subjects
* Subject will not be performing self-administration at home
* Does not transition to medication self-administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Change in patient-perceived medication knowledge and confidence. | Immediately before and after counseling session during 1 day study visit
  Patient knowledge and confidence will be assessed pre- and post-survey during the study counseling visit utilizing a modified Okere-Renier survey. Investigators hypothesize that patient knowledge and confidence in self-administering their biologic will increase after receipt of the combined nurse-pharmacist counseling intervention.

SECONDARY OUTCOMES:
Medication adverse events/self-administration errors | 90 days following study visit
  A pharmacist will perform a follow-up call at three months post-index. The pharmacist will interview the subject to determine if they experienced any ADEs or had any medication self-administration errors.
Medication adherence/persistence | 180 days following study visit
  Medication dispensing records for up to six months post-index at the study institution will be collected by extraction from pharmacy dispensing software by data manager. Medication adherence and persistence will be calculated in terms of PDC and discontinuation of the medication prior to 180 days.

CONTACTS AND LOCATIONS:
Overall Officials: Tonia Carr, BSN, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No